CLINICAL TRIAL: NCT02449655
Title: Trial of AZD5363 Plus Paclitaxel /AZD2014 Plus Paclitaxel in Biomarker Negative (PIK3CA/MEK/RAS/TP53/MET) Gastric Adenocarcinoma Patients as Second-line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of efficacy
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-04-122
Record Dates: First submitted 2015-05-14; First posted 2015-05-20 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — capivasertib; Paclitaxel; vistusertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD5363 plus paclitaxel (Experimental): AZD5363 4800mg bid 4 days on/ 3 days off of a 7 day cycle for each week that paclitaxel is given + paclitaxel 80mg/m2 given days 1, 8 and 15 of a 28 day cycle. AZD5363 and paclitaxel will be received for 3 consecutive weeks, followed by one week off-therapy in 4-week cycles.
  Interventions: Drug: AZD5363; Drug: paclitaxel
- AZD2014 plus paclitaxel (Active Comparator): AZD2014 50mg BD 3 days on 4 days off of a 7 day cycle + paclitaxel 80mg/m2 given days 1, 8 and 15 of a 28 day cycle
  Interventions: Drug: AZD2014; Drug: paclitaxel

INTERVENTIONS:
Drug: AZD5363 — AZD5363 4800mg bid 4 days on/ 3 days off of a 7 day cycle for each week
  Arms: AZD5363 plus paclitaxel
Drug: paclitaxel — paclitaxel 80mg/m2 given days 1, 8 and 15 of a 28 day cycle
  Arms: AZD5363 plus paclitaxel
Drug: AZD2014 — AZD2014 50mg BD 3 days on 4 days off of a 7 day cycle
  Arms: AZD2014 plus paclitaxel
Drug: paclitaxel — paclitaxel 80mg/m2 given days 1, 8 and 15 of a 28 day cycle
  Arms: AZD2014 plus paclitaxel

SUMMARY:
Phase II trial of AZD5363 plus paclitaxel / AZD2014 plus paclitaxel in biomarker negative (PIK3CA/MEK/RAS/TP53/MET) advanced gastric adenocarcinoma patients as second-line chemotherapy.

Each arm is composed of 25 patients.

AZD5363 400mg bid 4 days on/ 3 days off of a 7 day cycle for each week that paclitaxel is given + paclitaxel 80mg/m2 given days 1, 8 and 15 of a 28 day cycle. AZD5363 and paclitaxel will be received for 3 consecutive weeks, followed by one week off-therapy in 4-week cycles.If paclitaxel therapy is stopped then AZD5363 can be given on a 4on/3off continuous schedule.

AZD2014 50mg BD 3 days on 4 days off of a 7 day cycle + paclitaxel 80mg/m2 given days 1, 8 and 15 of a 28 day cycle.

Tumour evaluation using Response Evaluation Criteria in Solid Tumors 1.1 will be conducted at screening (within 28 days prior to first dose) and every 8 weeks relative to the date of first dose, up to week 40, then every 16 weeks until objective disease progression (within a window of +/- 7 days of the scheduled date).

Study treatment will be continued until objective disease progression.

The purpose of this study is to investigate the safety and efficacy of AZD5363 plus paclitaxel in biomarker negative (PIK3CA/MEK/RAS/TP53/MET) advanced gastric adenocarcinoma patients as second-line chemotherapy.

DETAILED DESCRIPTION:
AZD2014 is a selective dual mTOR kinase inhibitor targeting both mTORC1 (rapamycin sensitive) and mTORC2 (rapamycin insensitive) complexes of mammalian Target of Rapamycin (mTOR).

AZD2014 is a selective dual mTOR kinase inhibitor targeting both mTORC1 (rapamycin sensitive) and mTORC2 (rapamycin insensitive) complexes of mammalian Target Of Rapamycin (mTOR) AZD2014 is specific for mTOR and does not inhibit other members of the PI3K superfamily.

The PI3K-AKT-mTOR pathway functions as a sensor of mitogen, energy and nutrient levels and is a central controller of cell growth.

The mTOR is a protein kinase (PK) and a vital component of the PI3K/Akt/mTOR signaling pathway. This pathway is deregulated in 50% of all human cancers and, as such, is an important target for inhibitors that would alleviate the unregulated proliferation of cancer cells . AZD2014 is selective inhibitor of mTOR kinases and inhibits signalling of both mTOR complexes, mTORC1 and mTORC2.

In this study, the researchers further investigated the effect of PI3K/mTOR inhibitor as a paclitaxel sensitizer and/or nonspecific targeted therapy in combination with standard chemotherapy, paclitaxel in patients with pretreated advanced or metastatic gastric cancer having all negative biomarkers (PIK3CA/MEK/RAS/TP53/MET).

AZD5363 is a highly potent adenosine triphosphate (ATP)-competitive AKT inhibitor with IC50<10nmol/l for all three AKT isoforms.

AZD5363 is a highly potent adenosine triphosphate (ATP)-competitive AKT inhibitor with IC50<10nmol/l for all three AKT isoforms. AKT pathway is activated in various human cancers.Although AKT inhibitor has known showing anti-tumor activity in cell lines mutated at the E542, E545, or H1047 positions in preclinical study, clinical studies with AKT inhibitor are conducted for non-selected cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma that has progressed during or after first-line therapy.

   * The 1st line regimen must have contained doublet 5-fluoropyrimidine and platinum based regimen.
   * Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing doublet 5-fluoropyrimidine and platinum-based regimen could be considered as first line therapy.
4. Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the first line therapy.
5. Provision of tumor sample (from either a resection or biopsy)
6. Patients with biomarker negative
7. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
8. Eastern Cooperative Oncology Group performance status 0-1.
9. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
10. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥9.0 g/dL (transfusion allowed)
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * White blood cells (WBC) > 3 x 109/L
    * Platelet count ≥100 x 109/L (transfusion allowed)
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
    * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
    * Serum creatinine ≤1.5 x institutional ULN
11. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and following up visits.
12. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1.

Exclusion Criteria:

1. More than one prior chemotherapy regimen (except for adjuvant/neoadjuvant chemotherapy with more than 6 month wash out period) for the treatment of gastric cancer in the advanced setting.
2. Any previous treatment with PIK3CA, AKT or mTOR inhibitor or agents with mixed PI3K / mTOR activity.
3. Any previous treatment with paclitaxel
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
5. HER2 positive patients
6. Patients unable to swallow orally administered medication.
7. Any investigational drug or product administered within 30 days or 5 half-lives, whichever is longer, of the first dose of AZD5363.
8. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denusomab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
9. Previous major surgery within 4weeks prior to enrollment.
10. For AZD2014: Exposure to potent or moderate inhibitors or inducers of CYP3A4/5 if taken within the stated washout periods before the first dose of study treatment
11. With the exception of alopecia, any ongoing toxicities (>Common Toxicity Criteria for Adverse Effects grade 1) caused by previous cancer therapy.
12. Intestinal obstruction or Common Toxicity Criteria for Adverse Effects grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
13. Resting ECG with measurable QTcB > 480 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
14. Patients with cardiac problem as follows: uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) Left ventricular ejection fraction <55% measured by echocardiography, Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment
15. Active or untreated brain metastases or spinal cord compression Patients with treated brain metastases or spinal cord compression are eligible if they have minimal neurologic symptoms, evidence of stable disease (for at least 1 month) or response on follow-up scan, and require no corticosteroid therapy for ≥ 1 week.
16. Female patients who are breast-feeding or child-bearing
17. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)
18. Patients with proteinuria (3+ on dipstick analysis )

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | expected average of 24 weeks

SECONDARY OUTCOMES:
Duration of response | expected average of 24 weeks
Disease control rate | 8 weeks
Overall survival (OS) | expected average of 24 weeks
progression-free survival (PFS) | expected average of 24 weeks
Biomarker analysis | 3 years
  responders vs non-responders with whole exome sequencing/RNA sequencing including re-biopsy specimens Lauren classification (intestinal vs diffuse)
Number of subjects with Adverse Events as a measure of safety and tolerability | expected average of 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jee yun Lee, MD,Ph.D., Principal Investigator — Samsung Medical Center,Seoul,Korea
Locations (1):
- Samsung Medical center, Seoul, South Korea